CLINICAL TRIAL: NCT04900844
Title: A Multicenter, Single-Arm, Pivotal Study to Evaluate the Safety and Efficacy of the CGuard™ Carotid Stent System When Used to Treat Symptomatic and Asymptomatic Carotid Artery Stenosis in Patients Undergoing Carotid Artery Stenting
Brief Title: Safety and Efficacy of the CGuard™ Carotid Stent System in Carotid Artery Stenting
Acronym: C-Guardians
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: InspireMD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO-9017
Record Dates: First submitted 2021-05-20; First posted 2021-05-25 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Carotid Artery Stenosis
Keywords: Carotid Stenosis; Stenting; Prospective study; Embolic Protection Device (EPD); Carotid Artery Diseases; Cerebrovascular Disorders; Constriction, Pathologic
MeSH Terms: conditions — Carotid Stenosis; Carotid Artery Diseases; Cerebrovascular Disorders; Constriction, Pathologic

STUDY DESIGN:
Intervention Model Description: This is a single-arm trial, where the primary endpoint will be compared to a performance goal. The null hypothesis will be rejected (i.e. performance goal is met) if the upper bound of the two-sided 95% confidence interval calculated from the observed primary endpoint rate is < 11.6% and the p-value is less than 0.025.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- CGuard group (Experimental): Single experimental arm compared vs. objective performace goal
  Interventions: Device: CGuard Carotid Stent implantation

INTERVENTIONS:
Device: CGuard Carotid Stent implantation — Implantation of CGuard carotid stent in the eligible patients
  Other Names: Carotid stenting

SUMMARY:
The objective of this pivotal study is to evaluate the safety and efficacy of the CGuard™ Carotid Stent System in the treatment of carotid artery stenosis in symptomatic and asymptomatic patients undergoing carotid artery stenting (CAS) to a performance goal developed from published CAS literature.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is willing and able to provide appropriate study-specific informed consent, follow protocol procedures, and comply with follow-up visit requirements.
2. Subject is willing and able to take dual antiplatelet therapy for a minimum of 30 days.
3. Life expectancy ≥ 24 months from the date of the index procedure.
4. Females who are not pregnant or lactating and not planning to become pregnant for the duration of the study.
5. Subject has a modified Rankin Score of ≤ 2at the time of informed consent.
6. Subject is diagnosed with carotid artery disease treatable with carotid artery stenting and is considered high risk for carotid endarterectomy (CEA) as evidenced by:

   1. Symptomatic carotid stenosis ≥ 50%. Symptomatic is defined as amaurosis fugax, transient ischemia attack (TIA) or stroke within the last 6 months ipsilateral to the side of the stenosis.

      Or
   2. Asymptomatic carotid stenosis ≥ 80%
7. Co-Morbidity High Risk Conditions for CEA, i.e., meets one or more of the following criteria:

   1. Age ≥ 70 (maximum 80 years)
   2. CCS angina class 3-4 or unstable angina
   3. Congestive Heart Failure (CHF) NYHA class III-IV
   4. Left ventricular ejection fraction (LVEF) ≤ 35%
   5. MI ≥ 72 hours and < 6 weeks pre-procedure
   6. Multi-vessel CAD (≥ 2 vessels >70% stenosis) and history of angina
   7. Chronic Obstructive Pulmonary Disease (COPD) with FEV1<50
   8. Permanent contralateral cranial nerve injury/paralysis
   9. Restenosis from previous carotid endarterectomy (CEA)
   10. Planned coronary artery bypass grafting (CABG) or valve replacement surgery between 31-60 days after CAS
   11. Abdominal aortic aneurysm repair or peripheral vascular surgery is planned between 31 to 60 days after CAS.

   OR
8. High Anatomical Risk for CEA, i.e., meets one or more of the following criteria:

   1. Occlusion of the contralateral CCA or ICA.
   2. Prior radiation treatment to the neck or a radical neck dissection.
   3. Severe bilateral ICA stenosis requiring treatment.
   4. Target lesion at or above the level of the jaw (C2) or below the clavicle.
   5. Severe tandem lesions
   6. Inability to extend the hear due to cervical disorders.
   7. Laryngeal palsy or laryngectomy.
   8. Prior head and neck surgery in the region of the carotid artery.
   9. Tracheostomy or tracheostoma.
   10. Spinal immobility of the neck.
   11. Hostile neck or surgically inaccessible lesion.

10. Angiographic General Inclusion Criteria, i.e., meets all the following criteria:

1. Target lesion location at the carotid bifurcation and/or proximal internal carotid artery (ICA)
2. Vessel distal to target lesion can accommodate a distal embolic protection device (EPD), and EPD is compatible with CGuard™ device (refer to CGuard™ System IFU for specific EPDs).
3. Target vessel reference diameter at stent landing zone is 4.8 mm to 9.0 mm.
4. Target lesion length ≤ 36 mm, that can be covered by a single CGuard™ stent.

Exclusion Criteria:

1. Planned interventional procedure or surgery of the carotid, coronary or peripheral arteries within 30 days before or after the index carotid procedure.
2. Severe vascular anatomy that would preclude safe sheath insertion, deliverability of stent or embolic protection device.
3. Type III or bovine aortic arch.
4. Total occlusion of the target vessel.
5. Presence of "String sign" of the target lesion.
6. In-tandem lesions with >= 50% or >= 80% diameter stenosis for symptomatic or asymptomatic patients, respectively, which cannot be covered by a single CGuard™ stent.
7. History of bleeding diatheses or coagulopathy or inability to accept blood transfusions.
8. Bilateral carotid stenosis requiring treatment on both sides within 30 days prior to or following planned index procedure.
9. Subject is on renal replacement therapy or has Stage 4 or 5 Chronic Kidney Disease (CKD).
10. Known reason for potential stroke other than carotid artery stenosis, including history of atrial fibrillation or other sources of thromboemboli within the past 12 months.
11. History of thrombophilia.
12. Known sensitivity or allergy to nitinol, titanium, heparin, aspirin or other anticoagulant/ antiplatelet therapies.
13. Contrast media sensitivity or allergy that cannot be pre-treated.
14. Previous stent placement in the target vessel.
15. Evolving stroke or intracranial hemorrhage, or history of previous intracranial hemorrhage or brain surgery within the past 12 months.
16. Major neurologic deficit with NIHSS of ≥ 15.
17. Dementia or other neurologic condition confounding the neurologic assessment.
18. Clinical condition that, in the opinion of the investigator, makes endovascular therapy impossible or hazardous.
19. Subject previously enrolled in this clinical trial.
20. Possible / probable non-compliance of subject with protocol required follow up or medication.
21. Subject is currently participating in another clinical trial that has not completed its primary endpoint assessment or would confound this C-GUARDIANS Pivotal IDE Clinical Study.
22. SARS-CoV2 (COVID-19) active infection.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 317 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Composite of DSMI through 30 days or ipsilateral stroke 31 - 365 days post-index procedure | From index procedure to 1 year follow up
  The primary endpoint is the composite of the following:
  * Incidence of the following Major Adverse Events: Death (allcause mortality), all Stroke, and Myocardial Infarction (DSMI) through 30-days post-index procedure, based on Clinical Events Committee (CEC) adjudication OR
  * Ipsilateral stroke from 31-365 day follow-up, based on Clinical Events Committee (CEC) adjudication.

SECONDARY OUTCOMES:
Incidence of DSMI through discharge, 30 days, 6 months, and yearly follow ups till 3 years | From index procedure to 3 years follow up
  Incidence of the following composite of Major Adverse Events: Death (all-cause mortality), all Stroke, and Myocardial Infarction (DSMI) through discharge, 30-days, 6-months, and 1-,2-,3-year follow-up, based on Clinical Events Committee (CEC) adjudication.
Incidence of particular components of DSMI through discharge, 30 days, 6 months, and yearly follow ups till 3 years | From index procedure to 3 years follow up
  Incidence of each individual component of the Major Adverse Events: Death (all-cause mortality), all Stroke, and Myocardial Infarction (DSMI) through discharge, 30-days, 6-months, and 1-,2-,3-year follow-up, based on Clinical Events Committee (CEC) adjudication.
Incidence of ipsilateral stroke through discharge, 30 days, 6 months and 1-, 2-, 3-year follow-up. | From index procedure to 3 years follow up
  Ipsilateral stroke through discharge, 30 days, 6 months and 1-, 2-, 3-year follow-up.
Incidence of major ipsilateral stroke through discharge, 30 days, 6 months and 1-, 2-, 3-year follow-up. | From index procedure to 3 years follow up
  Major ipsilateral stroke through discharge, 30 days, 6 months and 1-, 2-, 3-year follow-up.
Incidence of In-stent Restenosis (ISR) > 70% in ultrasound evaluation | At 1-, 2-, 3-year post-index procedure follow-up
  Incidence of In-stent Restenosis (ISR) > 70%. ISR > 70% is defined as PSV > 300 cm/s associated with stent, or vessel occlusion based on transcervical duplex ultrasound through
  1-, 2-, 3-year follow-up. Based on Imaging Core Laboratory assessment.
Incidence of In-stent Restenosis (ISR) > 50% in ultrasound evaluation | At 1-, 2-, 3-year post-index procedure follow-up
  Incidence of In-stent Restenosis (ISR) > 50%. ISR > 50% is defined as PSV > 220 cm/s associated with stent, or vessel occlusion based on transcervical duplex ultrasound through
  1-, 2-, 3-year follow-up. Based on Imaging Core Laboratory assessment.
Incidence of target lesion revascularization | At 1-, 2-, 3-year post-index procedure follow-up
  Incidence of Target Lesion Revascularization (TLR) through 1-,2,3-year follow-up. TLR is defined as clinically driven revascularization procedure of the original treatment site, including angioplasty, stenting, endarterectomy, or thrombolysis, performed to open or increase the luminal diameter within the stented lesion or within 5 mm proximal or distal to the index stent.
Composite of Ipsilateral stroke, stent thrombosis, cardiovascular death or other device related clinical events | From index procedure to 3 years follow up
  Ipsilateral stroke, stent thrombosis, cardiovascular death or other device related clinical events from discharge up to 1-,2- and 3-year follow-up.
Composite of DSMI through 30 days or ipsilateral stroke 31 - 365 days post-index procedure for subjects that adhere to antiplatelet pharmacology. | From index procedure to 1 year follow up
  Primary endpoint for subjects that adhere to antiplatelet pharmacology.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Metzger, MD, Principal Investigator — Ballad Health; Piotr Musialek, MD DPhil, Principal Investigator — John Paul II Hospital, Krakow, Poland
Locations (18):
- United States (16):
  - University of Florida, Jacksonville, Florida
  - Oschner Health, New Orleans, Louisiana
  - Ascension, St. John Hospital, Detroit, Michigan
  - Mercy Hospital, St Louis, Missouri
  - University of Buffalo, Buffalo, New York
  - Columbia University Irving Medical Center, New York, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - Novant Health, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - UPMC-Pinnacle, Harrisburg, Pennsylvania
  - Miriam Hospital, Providence, Rhode Island
  - Prisma Health-Upstate, Greenville, South Carolina
  - Avera Heart Hospital, Sioux Falls, South Dakota
  - Ballad CVA Heart Institute, Kingsport, Tennessee
  - Turkey Creek Medical Center, Knoxville, Tennessee
  - Ascension Seton, Seton Heart Institute, Austin, Texas
- Poland (2):
  - Leszek Leic Upper-Silesian Medical Centre of the Silesian Medical University, Katowice
  - John Paul II Hospital, Krakow

IPD SHARING:
Plan to Share IPD: Yes